CLINICAL TRIAL: NCT05973617
Title: A Prospective Observational Study to Investigate the Role of the Biomechanics of the Cornea in Identifying Glaucoma or Anterior Eye Diseases and Create an IT Tool Able to Distinguish Between Them
Brief Title: Development of an IT Tool Able to Identify Ocular Conditions
Status: Withdrawn | Type: Observational
Why Stopped: Study did not commence
Sponsor: Aston University (Other)
Collaborators: Sandwell & West Birmingham Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 005-2021-SN
Record Dates: First submitted 2022-07-25; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Eye Diseases
Keywords: Machine Learning; Glaucoma; Keratoconus; Ocular Hypertension; Corneal Biomechanics
MeSH Terms: conditions — Eye Diseases; Glaucoma; Keratoconus; Ocular Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Glaucoma: Patients with diagnosis of glaucoma, that are receiving or had surgery to treat glaucoma
  Interventions: Diagnostic Test: Measurement of corneal biomechanical properties
- Ocular hypertension: Patients with diagnosis of ocular hypertension, that are receiving or had surgery to treat ocular hypertension
  Interventions: Diagnostic Test: Measurement of corneal biomechanical properties
- Keratoconus: Patients with diagnosis of keratoconus, that are receiving or had surgery to treat keratoconus
  Interventions: Diagnostic Test: Measurement of corneal biomechanical properties
- Healthy controls: Healthy
  Interventions: Diagnostic Test: Measurement of corneal biomechanical properties

INTERVENTIONS:
Diagnostic Test: Measurement of corneal biomechanical properties — Measurement of corneal biomechanics

SUMMARY:
The aim of the study is to use machine learning to develop an IT tool able to differentiate between eye conditions analysing corneal biomechanical data.

DETAILED DESCRIPTION:
Data will be collected using two different commercially available devices that are able to measure corneal biomechanics. Corneal biomechanics will be measured in participants with different conditions: glaucoma, ocular hypertension, corneal conditions, and healthy controls as it is well established that the above-mentioned conditions cause changes in corneal biomechanical properties.

Corneal biomechanics are the mechanical properties of the cornea, as rigidity, elasticity and it is possible to measure them using two devices: Ocular Response Analyzer (ORA) or Corneal Visualization Scheimpflug Technology (Corvis ST). Both devices use a puff of air to temporally flatten the cornea and derive the properties of the tissue.

Participants with ocular conditions will be recruited at Birmingham and Midlands Eye Centre (BMEC) at the Glaucoma and Anterior Eye clinics among patients attending for their routine clinical appointment. Healthy controls will be recruited at Aston University. This study requires only one visit and there is no need of follow up.

A portion of the data collected will be used to train machine learning algorithms to differentiate between conditions, the remaining data will be used to test the accuracy of newly created algorithms. The algorithm will be developed using Orange Data Mining.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years old.
* Participants who are able to give informed consent.
* Study groups: Patients with diagnosis of glaucoma or corneal disease or ocular hypertension. Patients that are having a treatment (medications or surgery) for glaucoma or ocular hypertension or corneal conditions.
* Control group: people with no diagnosis or treatment of previous pathologies.

Exclusion Criteria:

* Age below 18.
* Participants who are not able to give informed consent.
* Patients with eye conditions not within the inclusion criteria.
* Patients with respiratory distress or significant head tremor.
* Patients who are in pain or unable to remain seated for duration of measurements.
* Participants that during the visit are wearing contact lenses. The wear of contact lenses can alter the measure of corneal biomechanics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult population. Study group: patients at Birmingham and Midlands Eye Centre. Control groups: healthy population recruited in Birmingham among staff and students at Aston University.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
First applanation velocity | Day 1
  Velocity during the first applanation of the cornea, measured using Corivs ST [m/s]
First applanation time | Day 1
  Time frame of the first applanation of the cornea, measured using Corivs ST [s]
First applanation lenght | Day 1
  Lenght of the first applanation of the cornea, measured using Corivs ST [mm]
Second applanation velocity | Day 1
  Velocity during the second applanation of the cornea, measured using Corivs ST [m/s]
Second applanation time | Day 1
  Time frame of the second applanation of the cornea, measured using Corivs ST [s]
Second applanation lenght | Day 1
  Lenght of the second applanation of the cornea, measured using Corivs ST [mm]
Highest concavity time | Day 1
  Time frame at highest concavity, measured using Corivs ST [s]
Highest concavity peak distance | Day 1
  Distance between the 2 surrounding peaks at the highest concavity, measured using Corivs ST [mm]
Highest concavity radius | Day 1
  Radius of curvature at highest concavity, measured using Corivs ST [mm]
Highest concavity deformation amplitude | Day 1
  Maximal displacement of corneal apex between normal corneal shape and highest concavity, measured using Corivs ST [mm]
Corneal hysteresis | Day 1
  Difference in terms of intensity of puff of air between the first and second applanation, measured using ORA [mmHg]
Corneal resistance factor | Day 1
  Overall resistance of the cornea, measured using ORA [mmHg]

SECONDARY OUTCOMES:
Intraocular pressure measured using Corvis ST | Day 1
  Value of intraocular pressure measured according to the pressure of the air needed to applanate the cornea.
Intraocular pressure measured using ORA | Day 1
  Value of intraocular pressure measured according to the pressure of the air needed to applanate the cornea.
Pachymetry | Day 1
  Measure of corneal thickness using Corvis ST

CONTACTS AND LOCATIONS:
Overall Officials: Shehzad A Naroo, PhD, Principal Investigator — Aston University

IPD SHARING:
Plan to Share IPD: No